CLINICAL TRIAL: NCT06381856
Title: Improving Participation of Autistic Children and Adolescents in the Habilitation Process
Acronym: IMPAC
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: EPM_2024-00227-01
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism spectrum disorder; Patient participation; Needs assessment; Child; Adolescent; Parent
MeSH Terms: conditions — Autism Spectrum Disorder; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- survey based needs assessment: cohort receiving survey based needs assessment
- Personal meeting based assessment: cohort receiving personal meeting based needs assessment

SUMMARY:
This project aims to explore the impact of a survey-based and a meeting-based needs assessment models on 7 to 17 year old autistic children's participation in the needs assessment process at the initial reception when enrolled at a Child and Youth Habilitation Centre.

DETAILED DESCRIPTION:
The increasing number of children diagnosed with autism spectrum disorder (ASD) presents significant challenges for healthcare providers. Research emphasizes the importance of involving children in their healthcare decisions. However, due to the complex nature of ASD, characterized by differences in communication and social interaction, healthcare professionals struggle to adapt their services for these children.

To address this issue, the present study compares two assessment methods for children with ASD: one based on surveys and another based on meetings with healthcare professionals. In addition, supplementary information from the children's parents or guardians and healthcare providers will be gathered .

Data collection methods will include questionnaires, interviews, and analysis of individual habilitation plans. The goal is to recruit 120 children aged 7-17 diagnosed with ASD but without intellectual disabilities, with half undergoing the survey-based assessment and the other half undergoing the meeting-based assessment.

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum disorder

Exclusion Criteria:

* intellectual disability

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents receiving the survey based needs assessment and their parents/guardians (The survey-based needs assessment cohort).
  Children and adolescents receiving the personal meeting needs assessment and their parents/guardians (The personal-meeting needs assessment cohort).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The child's involvement | After each of four needs assessment meetings that take place over a 2-month period, with the first meeting scheduled to take place one month after inclusion.
  Consist of seven to nine questions relating to the child's involvement and engagement during a needs assessment meeting. The form is available in three versions. One for each child/youth, parent/guardian and staff. Each version comes in two variants. A variant for a regular meeting and a variant for the closing meeting. The questions are rated on 4-point Likert scales from "Not at all" to "Very much".

SECONDARY OUTCOMES:
The Mental Health Continuum - Short Form | At inclusion in the study and after completed needs assessment approximately 3 months after inclusion
  Consists of 14 questions which is assessed on a 6-point Likert scale and measures mental health in three domains (emotional, psychological and social well-being). The form appears in three versions. One where the child/youth assesses his/hers own health, one where the parent/guardian assesses his/hers own health and one where the parent/guardian assesses the child's/youth's health (i.e., proxy assessment).
The "Your child's strengths, abilities and special needs"-questionnaire. | At inclusion in the study and after completed needs assessment approximately 3 months after inclusion
  Consists of four or five questions from the "Family outcome survey" and adapted to the study's target group. The questions are answered by the parent/guardian and relate to their understanding of the child's strengths, abilities and special needs. The questions are answered on a 5-point scale Likert scales from "Nothing/Not at all" to "All/Always". The form is available in two variants. One for measurement before completed needs assessment (four questions) and one for measurement after completed needs assessment (five questions).
The collaboration with the neuropsychiatric team questionnaire | After completed needs assessment approximately 3 months after inclusion
  Consists of five questions relating to the family's contact with the neuropsychiatric team team at the Child and Youth Habilitation. The questions are answered with five answer options.
Cantril ladder | At inclusion in the study and after completed needs assessment approximately 3 months after inclusion
  Measures quality of life and is assessed on a picture of a ladder numbered from zero to ten.

OTHER OUTCOMES:
Individual interviews | After completed needs assessment, approximately 3 months after inclusion
  individual interviews with children, parents and healthcare professionals regarding how they experience the needs assessment procedure
Type and number of goals in the childrens' individual habilitation plans | After study completion, approximately 1 year after the start of the study.
  Type of goals described in the plans are categorized and the frequency of goals per category is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olov Lundqvist, Professor, Principal Investigator — Region Örebro County
Locations (1):
- University Health Care Research Center, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundqvist LO, Sjodin L, Karvonen E, Arnell S. Evaluating the impact of needs assessment models on autistic children's participation in the habilitation process: protocol for a prospective observational study. BMJ Open. 2024 Nov 1;14(10):e089135. doi: 10.1136/bmjopen-2024-089135. PMID 39486811